CLINICAL TRIAL: NCT01838941
Title: A Pilot, Open Label Trial Assessing the Safety and Efficacy of Betaine in Children With Peroxisome Biogenesis Disorders.
Brief Title: Betaine and Peroxisome Biogenesis Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Children's Hospital and Medical Center, Omaha, Nebraska (Other)
Responsible Party: Principal Investigator, Nancy Braverman, Associate Professor, Depts. of Human Genetics and Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPGDN001
Record Dates: First submitted 2013-03-29; First posted 2013-04-24 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Peroxisome Biogenesis Disorders
Keywords: Peroxisome Biogenesis Disorder; PBD; neonatal adrenoleukodystrophy; infantile Refsum disease; PEX1 mutation; Betaine
MeSH Terms: conditions — Peroxisome biogenesis disorders; Zellweger Syndrome; Peroxisomal Disorders; Refsum Disease, Infantile | interventions — Betaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Betaine (Experimental): Betaine will be given orally to all participants and dose will be adjusted to body weight.
  Interventions: Drug: Betaine

INTERVENTIONS:
Drug: Betaine — Betaine will be given orally (mixed with food or dissolved in water, juice, milk, or formula) or through gastrostomy tube as follows:
  * 6 g/day in children < 30 kg, in 3 divided doses (2 g at meal time)
  * 12 g/day in children > 30 kg, in 4 divided doses (3 g at meal time and bed time).
  Other Names: Cystadane®

SUMMARY:
The PBD are a rare group of inherited disorders due to the failure to form functional cellular peroxisomes. Most patients have progressive hearing and visual loss, leading to deafness and blindness, as well as neurological deterioration. There are no therapies for this disorder. A misfolded protein with residual function, PEX1-Gly843Asp, represents one third of all mutant alleles. Using patient cell lines with this mutation, we reported the recovery of peroxisome functions by treatment with Betaine, acting as a nonspecific chemical chaperone for the misfolded PEX1 protein. Betaine, or trimethylglycine, is a Health Canada and FDA approved orphan drug for the treatment of homocystinuria and is used by us safely and regularly in genetic medicine. We will perform a 6 month pilot study with 12 patients to test the hypothesis that Betaine, at recommended doses, can recover peroxisome biochemical functions in blood.

DETAILED DESCRIPTION:
Peroxisome biogenesis disorders (PBD) are a group of inherited conditions caused by faulty assembly of peroxisomes, structures located inside cells that regulate levels of important fats and lipids in the body. When there is faulty peroxisome assembly, as in PBD, these important fats and lipids either accumulate or are not made. There is no specific treatment for these disorders, and management is supportive. In order to complement existing supportive therapies, physicians and researchers are still actively looking for new treatments acting on the root cause of PBD: the peroxisome function. To identify drugs that help recover peroxisome function a group of scientists developed a laboratory-based research test aimed at reviewing the activity of the large number of potential treatments. Using this test, they have uncovered that Betaine can improve the function of the peroxisome, when the defect is caused by a PEX1-Gly843Asp mutation, and as such may improve the overall health of child suffering from PBD.

Betaine is a medication already available as a powder for oral solution, for another rare disease. It is approved in many countries, including Health Canada for Canada and the Food and Drug Administration for the USA. Paediatric genetic physicians are used to prescribing this medication and know it well.

At the current stage of scientific knowledge, it is a critical next step to evaluate the benefit of betaine in children having a PBD due to a PEX1-Gly843Asp mutation, to ensure that the medication is safe and to measure the level of improvement of the function of the peroxisome.

Thus, the principal objective of the study is to determine the improvement in the key peroxisome functions (plasma very long chain fatty acid profiles red cell plasmalogen levels, plasma pipecolic acid levels and plasma bile acid profiles). Another objective is to measure the growth of your child and his / her development.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* Any age
* Peroxisome Biogenesis Disorder (PBD) confirmed by biochemical analysis of at least two peroxisomal enzyme parameters:

  * Elevated plasma VLCFA (C26/22) > 0.02
  * Elevated plasma branched chain pristanic acid > 0.3 μg/ml
  * Reduced red blood cell plasmalogen levels (C16:0DMA/C16:0 Fatty acid) < 0.07
* PBD clinical syndromes: neonatal adrenoleukodystrophy (NALD) or infantile Refsum disease (IRD)
* Genotype PEX1-G843D/G843D, PEX1-G843D/I700fs, or PEX1-G843D and any second PEX1 mutation that is predicted to be null
* Expected survival of at least 6 months

Exclusion Criteria:

* Genotypes other than PEX1 G843D/G843D, PEX1-G843D//I700fs, or PEX1-G843D and any second PEX1 mutation that is predicted to be null
* Patient already treated with betaine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Braverman, PhD, MD, Principal Investigator — Montreal Children's Hospital, MUHC
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang R, Chen L, Jiralerspong S, Snowden A, Steinberg S, Braverman N. Recovery of PEX1-Gly843Asp peroxisome dysfunction by small-molecule compounds. Proc Natl Acad Sci U S A. 2010 Mar 23;107(12):5569-74. doi: 10.1073/pnas.0914960107. Epub 2010 Mar 8. PMID 20212125

RESULTS

PARTICIPANT FLOW:
Groups:
- Betaine: Betaine will be given orally to all participants and dose will be adjusted to body weight.
  Betaine: Betaine will be given orally (mixed with food or dissolved in water, juice, milk, or formula) or through gastrostomy tube as follows:
  * 6 g/day in children < 30 kg, in 3 divided doses (2 g at meal time)
  * 12 g/day in children > 30 kg, in 4 divided doses (3 g at meal time and bed time).
Period: Overall Study
Arm/Group | Betaine
Started | 12
Completed | 10
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Participants seen at research site; evaluation included physical examination, collection of medical history, measure of hematology, laboratory, and biochemical parameters.
Groups:
- Betaine: Betaine will be given orally to all participants and dose will be adjusted to body weight.
  Betaine: Betaine given orally (mixed with food or dissolved in water, juice, milk, or formula) or through gastrostomy tube:
  * 6 g/day in children < 30 kg, in 3 divided doses (2 g at meal time)
  * 12 g/day in children > 30 kg, in 4 divided doses (3 g at meal time and bed time).
Arm/Group | Betaine
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants] — Participants (n = 12) were seen at the research site at the beginning (baseline visit) and at the end of the study (6-month visit).
  Physical examination was done at baseline and final visits. Medical history was collected and updated at that time.
  Hematology, laboratory, and biochemical parameters were measured at baseline and 6 months.
  Participants
    <=18 years | 11
    Between 18 and 65 years | 1
    >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 4.75 [0.92 to 31.17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  Canada | 2
  United States | 10
Mutation status [Number; unit: participants] — Homozygous (mild form of PBD) or hemizygous for PEX1 G843D mutation (intermediate form of PBD)
  participants
    PEX1 G843D homozygous mutation | 2
    PEX1 G843D/null mutations | 10

OUTCOME MEASURES:

1. Primary Outcome: Peroxisome Biochemical Functions as Measured by Plasma Very Long Chain Fatty Acid
Description: C26/C22 ratio in plasma is a recognized biomarker for very long chain fatty acid (normal range: 0.002-0.018). It was measured twice before the beginning of treatment and measured once at the end.
Time Frame: 6 months
Measure: Mean (Full Range); unit: ratio
Groups:
- Betaine: Betaine will be given orally to all participants and dose will be adjusted to body weight.
  Betaine will be given orally (mixed with food or dissolved in water, juice, milk, or formula) or through gastrostomy tube as follows:
  * 6 g/day in children < 30 kg, in 3 divided doses (2 g at meal time)
  * 12 g/day in children > 30 kg, in 4 divided doses (3 g at meal time and bed time).
Arm/Group | Betaine
Number analyzed (Participants) | 10
ratio
  Baseline | 0.180 [0.027 to 0.301]
  At 6 months | 0.188 [0.059 to 0.286]

2. Secondary Outcome: Developmental Status
Description: Denver Developmental Screening Test expressed in years and months.
Time Frame: 6 months
Population: The Denver Developmental Screening Test was not performed.
Arm/Group | Betaine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Betaine
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Betaine (N=12)
Diarrhea (Gastrointestinal disorders) | 2 (3) — Diarrhea in 2 participants; duration: between 1 to 6 days.
Change in body odor (skin, urine, and/or breath) (Skin and subcutaneous tissue disorders) | 3 (4) — Change in breath in 2 participants; duration: up to 6 months Change in body odor (metallic smell) in 1 participant; duration: 2 months and a half. Change in urine odor in 2 participants; duration: 2 months.
Dry mouth (General disorders) | 1 (1) — Dry mouth in 1 participant; duration: 1 week.
Croup (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Croup in 1 participant; duration: 1 day.
Fatigue (General disorders) | 3 (3) — Fatigue in 3 participants; duration: 2 weeks to 4 months.
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Respiratory tract infection in 2 participants; duration: 7 to 10 days.
Gas (Gastrointestinal disorders) | 1 (1) — Gas in 1 participant; duration: 6 days.
Constipation (Gastrointestinal disorders) | 4 (4) — Constipation in 4 participants; duration: 6 to 9 days.
Vomiting (Gastrointestinal disorders) | 1 (1) — Vomiting in 1 participant; duration: 11 days.
Ear infection/Otitis media (Ear and labyrinth disorders) | 2 (9) — Ear infection/Otitis media in 2 participants; duration: 5 days to 1 month.
Increase in seizure activity (Nervous system disorders) | 1 (1) — Increase in seizure activity in 1 participant; duration: unknown
Decreased appetite (Gastrointestinal disorders) | 2 (2) — Decreased appetite in 2 participants; duration: up to 2 months
Upset stomach (Gastrointestinal disorders) | 1 (1) — Upset stomach in 1 participant; duration: 1 month
Viral syndrome (Infections and infestations) | 3 (4) — Viral syndrome in 3 participants; duration: approx. 5 days.
Elevated INR levels (Investigations) | 1 (1) — Elevated INR levels in 1 participant
Eye discharge (Eye disorders) | 1 (1) — Eye discharge in 1 participant.
Febrile seizure (Nervous system disorders) | 1 (2) — Febrile seizure in 1 participant; duration: 1 day

LIMITATIONS AND CAVEATS:
Large intra- and inter-individual variations in peroxisome functions, variation in phenotype severity, variation in age, number of participants; blood metabolite markers may be less sensitive than direct measurements of cell responses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No